CLINICAL TRIAL: NCT00400946
Title: Treatment of Acute Lymphoblastic Leukemia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lynda Vrooman, MD, Lynda Vroom, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-001 / CDR0000513019; P01CA068484 (NIH); P30CA006516 (NIH); DFCI-05001 (Other: DFCI IRB Protocol Number); NCT00165165 (obsolete NCT alias)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia
Keywords: drug/agent toxicity by tissue/organ; untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Dexamethasone; Dexrazoxane; Doxorubicin; Etoposide; Leucovorin; Mercaptopurine; Methotrexate; Methylprednisolone; pegaspargase; Prednisolone; Hydrocortisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramuscular native E coli L-asparaginase (IM-EC) (Active Comparator): Patients in this arm were randomized to intramuscular native E coli L-asparaginase 25 000 IU/m2 weekly for 30 doses. Protocol therapy was comprised of 5 phases: Induction, Consolidation I, CNS, Consolidation II, Continuation and varied dependent on risk classification. Patients who achieved complete remission after induction were eligible for post-induction asparaginase randomization. Further details are provided in the study description section.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: methylprednisolone; Drug: prednisolone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Intravenous PEG-asparaginase (IV-PEG) (Experimental): Patients in this arm were randomized to intravenous PEG-asparaginase 2500 IU/m2 every 2 weeks for 15 doses. Protocol therapy was comprised of 5 phases: Induction, Consolidation I, CNS, Consolidation II, Continuation and varied dependent on risk classification. Patients who achieved complete remission after induction were eligible for post-induction asparaginase randomization. Further details are provided in the study description section.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: methylprednisolone; Drug: pegaspargase; Drug: prednisolone; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: asparaginase
  Arms: Intramuscular native E coli L-asparaginase (IM-EC)
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: dexrazoxane hydrochloride
Drug: doxorubicin hydrochloride
Drug: etoposide — Given IV
Drug: leucovorin calcium
Drug: mercaptopurine — Given orally
Drug: methotrexate
Drug: methylprednisolone
Drug: pegaspargase — Given IV
  Arms: Intravenous PEG-asparaginase (IV-PEG)
Drug: prednisolone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: L-asparaginase is an important component of treatment for childhood acute lymphoblastic leukemia, but is also associated with notable side-effects, including hypersensitivity, pancreatitis, and thrombosis. We have previously reported that patients with acute lymphoblastic leukemia in whom asparaginase treatment was discontinued because of intolerable side-effects had survival outcomes that were inferior to those who received all or nearly all of their intended doses. Two bacterial sources of asparaginase exist: Escherichia coli (E coli) and Erwinia chrysanthemia (Erwinia). Generally, the E coli-derived enzyme has been used as front-line therapy and the Erwinia-derived preparation has been reserved for patients who develop hypersensitivity reactions. Pegylated E coli asparaginase (PEG-asparaginase) has a longer half-life and is potentially less immunogenic than native E coli L-asparaginase, and has been used as the initial asparaginase preparation in some pediatric acute lymphoblastic leukemia treatment regimens.

PURPOSE: Although the pharmacokinetics of each of these asparaginase preparations: intravenous PEG-asparaginase (IV-PEG) and intramuscular native E coli L-asparaginase (IM-EC) have been well characterized, their relative efficacy and toxicity have not been studied extensively.

DETAILED DESCRIPTION:
RISK CLASSIFICATION:

Patients received were classified into initial risk groups defined as:

High Risk (HR) High risk patients had any of the following features: age 10 years and older, a white blood cell count of 50 000 cells per μL or higher, initial spinal fluid sample with the presence of lymphoblasts and five or more white blood cells per high power field [Central Nervous System (CNS)-3], or a T-cell phenotype.

Standard Risk (SR) All other patients were classified as standard risk.

Patients who achieved complete remission (CR) after 32 days of induction therapy defined as a marrow specimen with less than 5% marrow blasts and evidence of normal haemopoiesis, absence of extramedullary disease, and recovery of peripheral blood counts were randomly assigned in a 1:1 ratio to receive IV-PEG or IM-EC. Randomization was stratified by final risk group assigned based on end-induction minimal residual disease and cytogenetics as follows:

Very High Risk (VHR)

Any initial risk group and any of the following:

* MLL gene rearrangement
* Hypodiploidy (<45 chromosomes)
* B cell-ALL (high) end-induction minimal residual disease (MRD) (>/= 0.001)

High Risk (HR)

No VHR features, plus:

HR initial risk group OR

SR initial risk group with either of the following:

* CNS-2 or CNS-3 on day 18
* CNS-2 on day 32 OR
* t(9;22) Philadelphia chromosome positive (Ph+ ALL)

Standard Risk (SR)

No VHR features, plus:

SR initial risk group AND

* CNS-1 on day 18 and 32

NOTE: CNS-1, Cerebral spinal fluid (CSF) without blasts; CNS-2, CSF with blasts and < 5 WBC per high-power field (HPF); CNS-3, CSF with blasts and ≥ 5 WBC per HPF

THERAPY:

INDUCTION

* Steroid prophase: Patients receive intrathecal (IT) cytarabine on day 1 and methylprednisolone IV every 8 hours on days 1-3. Patients then proceed to remission induction therapy.

Patients with CNS leukemia (CNS-2, CNS-3, or traumatic lumbar puncture [LP] with blasts) on initial LP receive additional IT cytarabine twice weekly beginning on days 4-6 and continuing until cerebrospinal fluid (CSF) is clear, followed by 2 additional doses. Patients with cranial nerve palsy but no leukemia blasts in CSF or leukemic eye infiltrates also receive additional IT cytarabine as above.

NOTE: Patients who received steroids within the past 7 days do not receive steroid prophase treatment; instead they proceed directly to remission induction therapy according to their risk group.

* Remission induction therapy (SR patients): Patients receive oral prednisone or prednisolone 2-3 times daily OR methylprednisolone IV every 8 hours on days 4-32; vincristine IV on days 4, 11, 18, and 25; doxorubicin hydrochloride (DOX) IV over 15 minutes on days 4 and 5; methotrexate (MTX) IV on day 6; pegasparaginase IV over 1 hour on day 7; triple intrathecal therapy (TIT) comprising methotrexate, cytarabine, and hydrocortisone on day 18; and IT MTX on day 32.
* Remission induction therapy (HR and VHR patients): Patients receive prednisone/prednisolone OR methylprednisolone; vincristine; DOX; MTX IV; pegasparaginase; TIT; and IT MTX as in the SR group. Patients also receive dexrazoxane hydrochloride IV over 15 minutes preceding the DOX infusions on days 4 and 5.

NOTE: Patients who do not receive steroid prophase treatment also receive IT cytarabine on day 4.

NOTE: Patients who are in CR on day 32 proceed to consolidation I. Patients who do not meet protocol definition of CR on day 32 but have no evidence of persistent disease receive vincristine IV weekly until CR is achieved. Patients with persistent marrow disease (greater than 5% leukemic blasts) and/or persistent extramedullary disease or those who do not achieve CR by day 53 are removed from the study.

NOTE: Patients with Ph+ ALL received imatinib (340 mg/m2 PO maximum 600 mg daily starting day 18) in combination with HR chemotherapy until they proceeded to stem cell transplant. Patients with Ph+ ALL patients did not participate in asparaginase randomization but were directly assigned to receive IM-EC during post-induction therapy.

CONSOLIDATION I

* Consolidation I (SR patients): Patients receive vincristine IV and IT MTX on day 1 and oral mercaptopurine once daily on days 1-14. Patients also receive high-dose MTX (HDM) IV continuously over 24 hours on day 1 and leucovorin calcium IV every 6 hours beginning 36 hours after the start of the HDM infusion and continuing until MTX levels are undetectable. Patients proceed to CNS therapy after day 21.
* Consolidation I (HR patients): Patients receive vincristine, IT MTX, and mercaptopurine as in the SR group. Patients also receive dexrazoxane hydrochloride IV over 15 minutes followed by DOX IV over 15 minutes on day 1 and HDM with leucovorin calcium support as in the SR group beginning 8-24 hours after the completion of the DOX infusion. Patients proceed to CNS therapy after day 21.
* Consolidation I (VHR patients): Patients receive consolidation therapy in 3 stages.

  * IA: Patients receive vincristine, IT MTX, and mercaptopurine as in the SR group. Patients also receive dexrazoxane hydrochloride, DOX, HDM, and leucovorin calcium as in the HR group.
  * IB: Patients receive cyclophosphamide IV over 1 hour and IT MTX on day 22; oral mercaptopurine once daily on days 22-35; and cytarabine IV on days 23-26 and 30-33.
  * IC: Patients receive high-dose cytarabine IV over 3 hours every 12 hours on days 43 and 44; etoposide IV over 1 hour on days 45-47; and oral dexamethasone twice daily on days 43-47. Patients also receive IM-EC weekly beginning on day 48 and continuing for up to 30 weeks OR IV-PEG over 1 hour every 2 weeks beginning on day 48 and continuing for up to 30 weeks. Patients proceed to CNS therapy after day 49.

KEY RANDOMIZATION: Patients are randomized 1:1 to receive either IV-PEG or IM-EC post-induction. Those who achieved a complete remission after induction therapy were assigned a final risk group and were eligible to participate in the randomization. The randomization was stratified by final risk group.

NOTE: Ph+ ALL patients did not participate in asparaginase randomization but were directly assigned to receive IM-EC during post-induction therapy. Patients who were eligible but declined randomization were also directly assigned to receive IM-EC. Patients who developed severe pancreatitis (defined as symptoms persisting for >72 h) during induction were not eligible for randomization and received no further doses of asparaginase. Patients who had hypersensitivity to IV-PEG during induction were also ineligible for randomization, but received twice-weekly IM-EC (25 000 IU/m2) during the post-induction treatment phases.

CNS

* CNS therapy (SR patients): Patients receive vincristine IV on day 1; oral mercaptopurine once daily on days 1-14; oral dexamethasone twice daily on days 1-5; and TIT twice weekly for 2 weeks. Patients also receive IV-PEG OR IM-EC as above beginning on day 1 and continuing for up to 30 weeks. Patients proceed to consolidation II after day 21.
* CNS therapy (HR and VHR patients): Patients receive vincristine, mercaptopurine, dexamethasone, and TIT as in the SR group. Patients also receive dexrazoxane hydrochloride IV over 15 minutes followed by DOX IV over 15 minutes on day 1. HR patients also receive IV-PEG OR IM-EC as above beginning on day 1 and continuing for up to 30 weeks. VHR patients continue to receive IV-PEG OR IM-EC as per consolidation I treatment. Patients proceed to consolidation II after day 21.

NOTE: Patients with WBC > 100,000/mm³, T-cell disease, and/or CNS-3 at diagnosis or CNS-2 at end of remission induction therapy also undergo cranial radiation therapy daily for 8 or 10 days.

CONSOLIDATION II

* Consolidation II (SR patients): Patients receive vincristine IV on day 1; oral dexamethasone twice daily on days 1-5; and oral mercaptopurine once daily on days 1-14. Treatment repeats every 21 days until IV-PEG OR IM-EC is completed. Patients also receive MTX IV or IM 1 day after each IV-PEG OR IM-EC dose and TIT every 9 weeks for 6 doses and then every 18 weeks thereafter.
* Consolidation II (HR and VHR patients): Patients receive vincristine, dexamethasone, and mercaptopurine as in the SR group. Patients also receive dexrazoxane hydrochloride IV over 15 minutes followed by DOX IV over 15 minutes on day 1. Treatment repeats every 21 days until IV-PEG OR IM-EC is completed. Patients also receive MTX IV or IM as in the SR group and TIT every 9 weeks for 6 doses and then every 18 weeks thereafter OR TIT every 18 weeks.

CONTINUATION

* Continuation therapy: After completion of all consolidation therapy, all patients receive vincristine IV on day 1; oral dexamethasone twice daily on days 1-5; oral mercaptopurine once daily on days 1-14; and MTX IV or IM on days 1, 8, and 15. Treatment repeats every 21 days for up to 24 months (102 weeks) after achieving CR. Patients continue to receive TIT as in consolidation II until completion of therapy.

OBJECTIVES:

Primary

* To determine the relative toxicity of IV PEG asparaginase and IM E.coli asparaginase in children with acute lymphoblastic leukemia (ALL)

Secondary (reported)

* To explore the relative efficacy of IV PEG asparaginase and IM E.coliasparaginase
* To determine the rate of infections (episodes of bacteremia and disseminated fungal infections) during the remission induction phase
* To compare trough serum asparaginase enzyme levels, asparagine levels and antiasparaginase antibody levels
* To evaluate the outcome of patients based upon MRD status after 28 days of multiagent chemotherapy within the context of a regimen which intensifies treatment for B-lineage patients with MRD levels >0.001 at the end of remission induction (day 32 MRD status used)
* To evaluate the outcome of patients based upon bone marrow morphology after 14 days of multiagent chemotherapy (day 18 marrow morphology status used)
* To determine the efficacy of CNS-directed treatments

Secondary (not reported)

* To compare antiasparaginase antibody levels (not available due to problems with the assay)
* To correlate trough enzyme levels with outcome (toxicity, relapse)
* To determine CNS-related toxicity of CNS-directed treatments (data is not mature on late neurocognitive impairments in long-term survivors)
* To determine the efficacy and CNS-related toxicity (acute and long-term) of the HR regimen in which a subset of HR patients (B-lineage, CNS-1 or CNS-2, WBC <100,000/m3) are treated with intensive intrathecal chemotherapy and the remainder are treated with 12 Gy cranial radiation (with intrathecal chemotherapy)
* To determine the efficacy and CNS-related toxicity (acute and long-term) of intensive intrathecal therapy in SR patients
* To determine the prognostic significance of asparaginase antibody formation
* To compare randomized treatment groups using health-related quality-of-life analysis (connected with a separate protocol 06-373)
* To investigate the association of dietary antioxidant micronutrient intake with the rate of infections (episodes of bacteremia and disseminated fungal infections) during remission induction therapy and the Consolidation IA phase
* To determine the relationship of dietary calcium intake with risk for development of fractures during the continuation phase of therapy
* To evaluate the association of dietary intake of specific nutrients with treatment-related toxicities during treatment
* To evaluate the outcome of patients based upon MRD status after 14 days of multiagent chemotherapy and at various other timepoints while on treatment every 18 weeks after achieving complete remission and at the completion of all chemotherapy
* To determine the prognostic significance of response to remission induction chemotherapy as measured by morphologic and minimal residual disease (MRD) measures within the context of DFCI ALL Consortium protocol therapy (data limited due to response outcomes)
* To compare rate of infection during remission induction in patients treated with a less intensive induction regimen on Protocol 05-01 (low-dose instead of high-dose methotrexate) with that of patients treated on prior DFCI ALL Consortium Protocol 00-01 (induction regimen included high-dose methotrexate)
* To determine the concordance of MRD quantification using multi-parameter flow cytometry and PCR techniques
* To determine the prognostic significance of gene expression programs in childhood ALL and identify new targets for specific therapies
* To identify clinically relevant gene expression signatures in leukemia cells
* To identify gene expression signature in leukemia cells at diagnosis that predicts peripheral blood response to the steroid prophase
* To identify gene expression changes in leukemia cells induced by steroid treatment
* To determine the frequency and type of tyrosine kinase mutations in childhood ALL and identify new targets for specific therapies
* To explore the potential relationship between abnormal glucose homeostasis during therapy and the development of obesity, as well as the potential relationship between obesity and the age of pubertal onset (assessed in patients treated at DFCI/CHB only)
* To characterize the degree of hyperglycemia and insulin resistance in patients receiving therapy for childhood ALL
* To characterize the degree of insulin resistance and obesity after the completion of therapy for childhood ALL

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * No known mature B-cell ALL, defined by the presence of any of the following:

    * Surface immunoglobulin
    * L3 morphology
    * t(8;14)(q24;q32)
    * t(8;22)
    * t(2;8)
  * T-cell surface markers and t(8;14)(q24;q11) allowed
* No secondary ALL

PATIENT CHARACTERISTICS:

* No known HIV positivity
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior therapy except steroids of ≤ 1 week in duration and/or emergent radiation therapy to the mediastinum

  * Patients treated with steroids within the past 7 days will not receive steroid prophase during study treatment

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Vrooman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Hasbro Children's Hospital, Providence, Rhode Island
- Canada (3):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silverman LB, Supko JG, Stevenson KE, Woodward C, Vrooman LM, Neuberg DS, Asselin BL, Athale UH, Clavell L, Cole PD, Kelly KM, Laverdiere C, Michon B, Schorin M, Schwartz CL, O'Brien JE, Cohen HJ, Sallan SE. Intravenous PEG-asparaginase during remission induction in children and adolescents with newly diagnosed acute lymphoblastic leukemia. Blood. 2010 Feb 18;115(7):1351-3. doi: 10.1182/blood-2009-09-245951. Epub 2009 Dec 10. PMID 20007809
- [Result] Place AE, Stevenson KE, Vrooman LM, Harris MH, Hunt SK, O'Brien JE, Supko JG, Asselin BL, Athale UH, Clavell LA, Cole PD, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Schorin MA, Welch JJ, Lipshultz SE, Kutok JL, Blonquist TM, Neuberg DS, Sallan SE, Silverman LB. Intravenous pegylated asparaginase versus intramuscular native Escherichia coli L-asparaginase in newly diagnosed childhood acute lymphoblastic leukaemia (DFCI 05-001): a randomised, open-label phase 3 trial. Lancet Oncol. 2015 Dec;16(16):1677-90. doi: 10.1016/S1470-2045(15)00363-0. Epub 2015 Nov 6. PMID 26549586
- [Derived] Vrooman LM, Blonquist TM, Harris MH, Stevenson KE, Place AE, Hunt SK, O'Brien JE, Asselin BL, Athale UH, Clavell LA, Cole PD, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Schorin MA, Sulis ML, Welch JJG, Neuberg DS, Sallan SE, Silverman LB. Refining risk classification in childhood B acute lymphoblastic leukemia: results of DFCI ALL Consortium Protocol 05-001. Blood Adv. 2018 Jun 26;2(12):1449-1458. doi: 10.1182/bloodadvances.2018016584. PMID 29941458
- [Derived] Kahn JM, Cole PD, Blonquist TM, Stevenson K, Jin Z, Barrera S, Davila R, Roberts E, Neuberg DS, Athale UH, Clavell LA, Laverdiere C, Leclerc JM, Michon B, Schorin MA, Welch JJG, Sallan SE, Silverman LB, Kelly KM. An investigation of toxicities and survival in Hispanic children and adolescents with ALL: Results from the Dana-Farber Cancer Institute ALL Consortium protocol 05-001. Pediatr Blood Cancer. 2018 Mar;65(3):10.1002/pbc.26871. doi: 10.1002/pbc.26871. Epub 2017 Nov 1. PMID 29090520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from April 22, 2005 to Dec 13, 2011.
Groups:
- IM-EC [Directly Assigned]: Ph+ ALL patients did not participate in asparaginase randomization but were directly assigned to receive intramuscular E coli L-asparaginase during post-induction therapy. Patients who were eligible but declined randomization were also directly assigned to receive intramuscular E coli L-asparaginase.
- Ineligible for Randomization: All patients received a single dose of intravenous PEG-asparaginase 2500 IU/m2 during multi-agent induction. Patients who did not achieve complete remission and were not assigned a final risk group by the end of the induction phase of treatment were not eligible for randomization. Patients who developed severe pancreatitis (defined as symptoms persisting for >72 h) during induction were not eligible for randomization and received no further doses of asparaginase. Patients who had hypersensitivity to intravenous PEG-asparaginase during induction were also ineligible for randomization, but received twice-weekly IM-EC (25 000 IU/m2) during the post-induction treatment phases.
- Expansion Cohort: Patients were enrolled in an expansion cohort to determine the prognostic significance of response to remission induction chemotherapy as measured by morphologic and minimal residual disease (MRD), and to further evaluate the efficacy of patients by final risk classification.
Period: Overall Study
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG) | IM-EC [Directly Assigned] | Ineligible for Randomization | Expansion Cohort
Started | 231 | 232 | 42 | 51 | 244
Evaluable for CNS Directed-Treatment (Patients who achieved an induction complete remission with an evaluable sample at diagnosis.) | 231 | 232 | 42 | 21 | 227
Evaluable for Day 18 Marrow Morphology (Patients who achieved an induction complete remission with an optional evaluable sample at day 18.) | 158 | 161 | 19 | 13 | 152
Evaluable for Day 32 MRD (B cell patients who achieved an induction complete remission with an evaluable sample at day 32.) | 166 | 167 | 33 | 12 | 168
Eligible and Treated (Ineligible: Burkitt's leuk diag (n=2), pr therapy (n=1), hyperbilirubinemia (n=1), w/d consent (n=2)) | 231 | 232 | 42 | 46 | 243
Completed | 217 | 221 | 40 | 4 | 206
Not Completed | 14 | 11 | 2 | 47 | 38
Not completed — Ineligible | 0 | 0 | 0 | 5 | 1
Not completed — Induction Failure | 0 | 0 | 0 | 11 | 8
Not completed — Induction Death | 0 | 0 | 0 | 13 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1
Not completed — Remission Death | 1 | 1 | 0 | 0 | 1
Not completed — Relapse | 9 | 2 | 1 | 1 | 5
Not completed — Transplant in CR1 | 0 | 0 | 0 | 10 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 1 | 5 | 8
Not completed — Clinical | 1 | 2 | 0 | 2 | 9
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG) | IM-EC [Directly Assigned] | Ineligible for Randomization | Expansion Cohort | Total
Number analyzed (Participants) | 231 | 232 | 42 | 51 | 244 | 800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 231 | 232 | 42 | 51 | 244 | 800
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 97 | 21 | 21 | 107 | 357
  Male | 120 | 135 | 21 | 30 | 137 | 443
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 48 | 3 | 13 | 48 | 152
  Not Hispanic or Latino | 165 | 170 | 35 | 34 | 180 | 584
  Unknown or Not Reported | 26 | 14 | 4 | 4 | 16 | 64
Age Classification [Count of Participants; unit: Participants]
  < 10 years old | 176 | 165 | 35 | 26 | 196 | 598
  >/= 10 years old | 55 | 67 | 7 | 25 | 48 | 202

OUTCOME MEASURES:

1. Primary Outcome: Asparaginase-Related Toxicity Rate
Description: Asparaginase-related toxicity rate is defined as the percentage of patients who experience allergy (all grades), symptomatic pancreatitis (grade 2 or worse), thrombotic or bleeding complications requiring intervention (grade 2 or worse) with treatment attribution of possibly, probably or definite based on CTCAEv3.
Time Frame: 30-week post-induction asparaginase treatment period
Population: The analysis dataset is comprised of all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG)
Number analyzed (Participants) | 231 | 232
percentage of participants | 26 [20 to 32] | 28 [22 to 34]
Statistical Analysis 1: Comparison: Intramuscular Native E Coli L-asparaginase (IM-EC) vs Intravenous PEG-asparaginase (IV-PEG); Test type: Superiority; p = .60, Fisher Exact

2. Secondary Outcome: 5-Year Disease-Free Survival
Description: Disease-free survival (DFS) in a landmark analysis is defined as the duration of time from asparaginase randomization (which occurred after patients achieved complete remission and were assigned to a final risk group) to documented relapse, death during remission or second malignant neoplasm. DFS is estimated based on the Kaplan-Meier method and 5-year DFS is the probability of patients remaining alive, relapse-free and without occurrence of second malignant neoplasm 5 years from asparaginase randomization. Disease relapse is defined as >25% lymphoblasts identified morphologically in bone marrow aspirate/biopsy, or identification of lymphoblasts in marrow (any percentage) identified to be leukemic by flow cytometry, cytogenetics, FISH, immunohistochemistry, or other tests. Appearance of leukemic cells at any extramedullary site (a single, unequivocal lymphoblast in the CSF may qualify as CNS leukemia) also qualifies if confirmed by the PI.
Time Frame: Disease evaluations occurred continuously on treatment. Suggested long-term follow-up was monthly for 6m, bi-monthly for 6m, every 4 months for 1y, semi-annually for 1y, then annually. Median follow-up in this study cohort is 6 yrs, up to 10y.
Population: The analysis dataset is comprised of all randomized patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG)
Number analyzed (Participants) | 231 | 232
probability | .89 [.85 to .93] | .90 [.86 to .94]

3. Secondary Outcome: Post-Induction Nadir Serum Asparaginase Activity Level
Description: Nadir serum asparaginase activity (NSAA) levels were estimated based on established methods.
Time Frame: Samples for nadir serum asparaginase activity analyses were obtained before doses administered at weeks 5, 11, 17, 23 and 29 of post-induction asparaginase treatment.
Population: The analysis dataset is comprised of all randomized patients who consented to research studies with an evaluable sample for analysis of serum asparaginase activity at the respective post-induction assessment timepoints.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG)
Number analyzed (Participants) | 231 | 232
IU/mL
  Week 5 NSAA Level: number analyzed (Participants) | 76 | 78
  Week 5 NSAA Level | 0.129 (0.108) | 0.726 (0.322)
  Week 11 NSAA Level: number analyzed (Participants) | 69 | 76
  Week 11 NSAA Level | 0.143 (0.131) | 0.773 (0.231)
  Week 17 NSAA Level: number analyzed (Participants) | 85 | 80
  Week 17 NSAA Level | 0.159 (0.161) | 0.787 (0.303)
  Week 23 NSAA Level: number analyzed (Participants) | 75 | 66
  Week 23 NSAA Level | 0.180 (0.261) | 0.757 (0.255)
  Week 29 NSAA Level: number analyzed (Participants) | 53 | 69
  Week 29 NSAA Level | 0.123 (0.102) | 0.806 (0.313)

4. Secondary Outcome: Post-Induction Therapeutic Nadir Serum Asparaginase Activity Rate
Description: Nadir serum asparaginase activity (NSAA) levels were estimated based on established methods. Post-Induction therapeutic NSAA rate is defined as the percentage of patients achieving a NSAA level above 0.1 IU/mL ever during post-induction therapy.
Time Frame: as for outcome 3
Population: The analysis dataset is comprised of all randomized patients who consented to research studies with a one post-induction evaluable sample for analysis of serum asparaginase activity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG)
Number analyzed (Participants) | 170 | 168
percentage of participants | 71 [63 to 77] | 99 [96 to 99]

5. Secondary Outcome: Induction Infection Toxicity Rate
Description: Infection toxicity rate is defined as the percentage of patients who experience bacterial or fungal infection of grade 3 or higher with treatment attribution of possibly, probably or definite based on CTCAEv3 during remission induction phase of combination chemotherapy.
Time Frame: Assessed daily during remission induction days 4-32.
Population: The analysis dataset is comprised of eligible and treated patients. This excludes the 6 enrolled but ineligible patients. Rates in this overall study cohort will be compared against historical controls (in particular patients treated with a more intensive induction regimen).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall: Protocol therapy was comprised of 5 phases: Induction, Consolidation I, CNS, Consolidation II, Continuation and varied dependent on risk classification. All patients received a single dose of intravenous PEG-asparaginase 2500 IU/m2 during multi-agent induction. Patients who achieved complete remission after induction were eligible for post-induction asparaginase randomization wherein patients received either E. coli L-asparaginase or peg-asparaginase. Standard risk and high-risk patients began post-induction randomized asparaginase therapy at the start of the CNS phase, whereas very high-risk patients began asparaginase therapy on day 8 of consolidation phase IC. Patients who did not achieve complete remission by the end of the induction phase were not eligible for randomization, were removed from protocol treatment, and received alternative therapy according to the discretion of their treating physician. Further details are provided in the study description section.
Arm/Group | Overall
Number analyzed (Participants) | 794
percentage of participants | 26 [23 to 30]

6. Secondary Outcome: Induction Serum Asparaginase Activity Level
Description: Serum asparaginase activity (NSAA) levels were estimated based on established methods.
Time Frame: Samples for serum asparaginase activity analyses were obtained days 4, 11, 18 and 25 post one-dose of IV-PEG on day 7 of the induction phase.
Population: The analysis dataset is comprised of all randomized patients who consented to research studies with an evaluable sample for analysis of serum asparaginase activity at the respective induction assessment timepoints.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Overall
Number analyzed (Participants) | 794
IU/mL
  Day 4 NSAA Level: number analyzed (Participants) | 317
  Day 4 NSAA Level | .694 [.556 to .868]
  Day 11 NSAA Level: number analyzed (Participants) | 348
  Day 11 NSAA Level | .505 [.306 to .632]
  Day 18 NSAA Level: number analyzed (Participants) | 294
  Day 18 NSAA Level | .211 [.150 to .259]
  Day 25 NSAA Level: number analyzed (Participants) | 298
  Day 25 NSAA Level | .048 [.025 to .076]

7. Secondary Outcome: Induction Therapeutic Nadir Serum Asparaginase Activity Rate
Description: Nadir serum asparaginase activity (NSAA) levels were estimated based on established methods. Induction therapeutic NSAA rate is defined as the percentage of patients achieving a NSAA level above 0.1 IU/mL at a given timepoint.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Overall
Number analyzed (Participants) | 794
percentage of participants
  Day 4 NSAA Rate: number analyzed (Participants) | 317
  Day 4 NSAA Rate | 97
  Day 11 NSAA Rate: number analyzed (Participants) | 348
  Day 11 NSAA Rate | 96
  Day 18 NSAA Rate: number analyzed (Participants) | 294
  Day 18 NSAA Rate | 87
  Day 25 NSAA Rate: number analyzed (Participants) | 298
  Day 25 NSAA Rate | 12

8. Secondary Outcome: 5-Year Disease-Free Survival by MRD Day 32 Status
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of B cell ALL patients who achieved an induction complete remission with an evaluable sample at day 32 for analysis of MRD.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Low Day 32 MRD Level: Low end-induction (day 32) minimal residual disease (MRD) evaluated was defined as <0.001. This MRD classification was one component of determining final risk classification. Peripheral blood samples were collected for evaluation of MRD using PCR methods.
- High Day 32 MRD Level: High end-induction (day 32) minimal residual disease (MRD) evaluated was defined as >/=0.001. This MRD classification was one component of determining final risk classification. Peripheral blood samples were collected for evaluation of MRD using PCR methods
Arm/Group | Low Day 32 MRD Level | High Day 32 MRD Level
Number analyzed (Participants) | 50 | 496
probability | .79 [.60 to .86] | .90 [.87 to .93]

9. Secondary Outcome: 5-Year Disease-Free Survival by Bone Marrow Day 18 Status
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of patients who achieved an induction complete remission with an evaluable sample at day 18 (optional submission) for analysis of marrow morphology.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- M1 Day 18 Bone Marrow Status: M1 marrow morphology at day 18 was defined as <5% blasts.
- M2/M3 Day 18 Bone Marrow Status: M2 marrow morphology at day 18 was defined as 5-24% blasts. M3 marrow morphology at day 18 was defined as >25% blasts.
- Hypocellular Day 18 Bone Marrow Status: Hypocellular marrow morphology at day 18 was defined as empty blasts.
Arm/Group | M1 Day 18 Bone Marrow Status | M2/M3 Day 18 Bone Marrow Status | Hypocellular Day 18 Bone Marrow Status
Number analyzed (Participants) | 284 | 26 | 193
probability | .89 [.85 to .92] | .78 [.54 to .90] | .88 [.82 to .92]

10. Secondary Outcome: 5-year Disease-Free Survival by CNS Directed Treatment Group
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of patients who achieved an induction complete remission with an evaluable sample at diagnosis for analysis of CNS-directed therapy .
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- CNS-1: CNS-1: no blast cells in cytospin, regardless of cerebrospinal fluid (CSF) count
- CNS-2: CNS-2: 5 or fewer WBC on CSF cell count, with blasts on cytospin
- CNS-3: CNS-3: more than 5 WBC on CSF cell count, with blasts on cytospin
- Traumatic Tap With Blasts: Traumatic Tap with Blasts: with blast cells and >100 RBCs on a wet prep
- Traumatic Tap Without Blasts: Traumatic Tap without Blasts: without blast cells and >100 RBCs on a wet prep
Arm/Group | CNS-1 | CNS-2 | CNS-3 | Traumatic Tap With Blasts | Traumatic Tap Without Blasts
Number analyzed (Participants) | 579 | 114 | 9 | 32 | 19
probability | .89 [.87 to .92] | .89 [.82 to .94] | 1.00 [NA to NA] — NA-not applicable since all patients were disease-free at 5 years. | .84 [.67 to .93] | .87 [.58 to .97]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were continuously monitored and reported every 3 months during treatment except bony events (avascular necrosis and fracture) which were followed up to 10 years. Treatment duration for this study cohort was a median (range) of 757 days (1-881 days). Data is reported for the entire study cohort (n=794) and comparing randomized arms (n=231/n=232), other non-randomized reporting groups are not reported separately since the intent was not to compare rates between these groups.
Description: Reporting included (trt-related, all grades [G] unless specified): asparaginase-related allergy, symptomatic pancreatitis (>G1), thrombotic or bleeding complications requiring intervention (>G1), infections (>G2), symptomatic osteonecrosis (>G1), bone fractures and seizures. All other G4-5 AEs were also collected, excl G4 hematological and G4 asymptomatic elevated aminotransferases. Maximum grade toxicity by type was calculated with serious and other AEs defined as G3-5 and G1-2, respectively.
Arm/Group | Intramuscular Native E Coli L-asparaginase (IM-EC) | Intravenous PEG-asparaginase (IV-PEG) | Overall
All-Cause Mortality (participants affected / at risk) | 1/231 | 1/232 | 2/794
Serious Adverse Events (participants affected / at risk) | 132/231 | 142/232 | 574/794
Other Adverse Events (participants affected / at risk) | 40/231 | 38/232 | 118/794
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intramuscular Native E Coli L-asparaginase (IM-EC) (N=231) | Intravenous PEG-asparaginase (IV-PEG) (N=232) | Overall (N=794)
Acute vascular leak syndrome (Vascular disorders) | 0 | 0 | 1
ADH secretion abnormality (eg SIADH) (Investigations) | 0 | 0 | 1
Alkaline phosphatase (Investigations) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bronchopulmonary- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cardiac-other (Cardiac disorders) | 0 | 0 | 1
Cecum/appendix- hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chyle or lymph leakage (Vascular disorders) | 0 | 1 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 1
Coagulation-other (Investigations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Creatinine (Investigations) | 0 | 0 | 1
Death - multiorgan failure (General disorders) | 0 | 0 | 1
Death - sudden death (General disorders) | 0 | 0 | 1
Edema limb (General disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Head/headache (Nervous system disorders) | 0 | 0 | 1
Hematologic-other (Blood and lymphatic system disorders) | 0 | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Infection Gr0-2 neut- bladder (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- bronchus (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut- cervix (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- dental-tooth (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut- middle ear (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- muscle (Infections and infestations) | 0 | 1 | 1
Infection Gr0-2 neut- soft tissue (Infections and infestations) | 0 | 1 | 1
Infection Gr0-2 neut- spleen (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- brain (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- brain + spinal (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- dental-tooth (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- eye NOS (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- lens (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- lip/perioral (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- liver (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- paranasal (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- pleura (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- sinus (Infections and infestations) | 1 | 0 | 1
Infection w/ gr3-4 neut- spinal cord (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- spleen (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- trachea (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- vein (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC abdomen NOS (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC colon (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC lymphatic (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC meninges (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 0 | 1
INR (Investigations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Intra-op injury Other (Specify) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intra-op injury Pleura (Injury, poisoning and procedural complications) | 1 | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 1 | 1
Joint- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Kidney- pain (Renal and urinary disorders) | 0 | 1 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 0 | 1 | 1
Lung- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Necrosis- pancreas (Gastrointestinal disorders) | 0 | 1 | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Obstruction-ureteral (Renal and urinary disorders) | 0 | 0 | 1
Oral cavity- pain (Gastrointestinal disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain NOS (General disorders) | 0 | 1 | 1
Pelvic- pain (Reproductive system and breast disorders) | 0 | 0 | 1
Perforation- appendix (Renal and urinary disorders) | 0 | 0 | 1
Perforation- stomach (Gastrointestinal disorders) | 0 | 1 | 1
Peripheral arterial ischemia (Vascular disorders) | 0 | 1 | 1
Personality (Psychiatric disorders) | 0 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PTT (Investigations) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Soft tissue necrosis- extremity lower (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 0 | 1
Surgical hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Ulcer- anus (Gastrointestinal disorders) | 0 | 0 | 1
Ulcer- duodenum (Gastrointestinal disorders) | 0 | 0 | 1
Ulcer- esophagus (Gastrointestinal disorders) | 0 | 0 | 1
Ulcer- gastric (Gastrointestinal disorders) | 0 | 1 | 1
Urinary electrolyte wasting (Metabolism and nutrition disorders) | 1 | 0 | 1
Varices (esophageal)- hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 2 | 2
Bone- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 2
Confusion (Psychiatric disorders) | 1 | 0 | 2
Duodenum- hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 2
Fever w/o neutropenia (General disorders) | 0 | 1 | 2
Hypercholesterolemia (Investigations) | 0 | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Infection Gr0-2 neut- abdomen (Infections and infestations) | 0 | 1 | 2
Infection Gr0-2 neut- catheter (Infections and infestations) | 0 | 1 | 2
Infection Gr0-2 neut- eye NOS (Infections and infestations) | 0 | 1 | 2
Infection Gr0-2 neut- liver (Infections and infestations) | 0 | 0 | 2
Infection Gr0-2 neut- peritoneal (Infections and infestations) | 0 | 0 | 2
Infection Gr0-2 neut- wound (Infections and infestations) | 2 | 0 | 2
Infection w/ gr3-4 neut- anal/perianal (Infections and infestations) | 0 | 0 | 2
Infection w/ gr3-4 neut- kidney (Infections and infestations) | 0 | 1 | 2
Infection w/ gr3-4 neut- meninges (Infections and infestations) | 0 | 0 | 2
Infection w/ gr3-4 neut- middle ear (Infections and infestations) | 1 | 0 | 2
Infection w/ gr3-4 neut- peritoneal (Infections and infestations) | 0 | 0 | 2
Infection w/ gr3-4 neut- urinary tract (Infections and infestations) | 1 | 0 | 2
Infection w/ unk ANC bladder (Infections and infestations) | 0 | 0 | 2
Infection w/ unk ANC lung (Infections and infestations) | 0 | 0 | 2
Infection w/ unk ANC wound (Infections and infestations) | 0 | 0 | 2
Lower GI- hemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | 2
Oral gums- pain (Gastrointestinal disorders) | 1 | 1 | 2
Pain-other (General disorders) | 1 | 0 | 2
Perforation- small bowel NOS (Gastrointestinal disorders) | 0 | 1 | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 3
Depression (Psychiatric disorders) | 1 | 1 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 0 | 3
Fibrinogen (Investigations) | 0 | 0 | 3
Leukocytes (Investigations) | 0 | 0 | 3
Myelitis (Nervous system disorders) | 0 | 1 | 3
Neurologic-other (Nervous system disorders) | 1 | 1 | 3
Psychosis (Psychiatric disorders) | 0 | 1 | 3
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Skin-other (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Upper GI- hemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 3
Abdomen- pain (Gastrointestinal disorders) | 0 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 4
Ileus (Gastrointestinal disorders) | 0 | 0 | 4
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 2 | 0 | 4
Infection w/ gr3-4 neut- catheter relate (Infections and infestations) | 0 | 0 | 4
Infection w/ gr3-4 neut- upper airway (Infections and infestations) | 2 | 1 | 4
Infection w/ gr3-4 neut- wound (Infections and infestations) | 0 | 1 | 4
Metabolic/Laboratory-other (Investigations) | 0 | 1 | 4
Neuropathy-sensory (Nervous system disorders) | 2 | 0 | 4
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 4
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
CNS- hemorrhage (Nervous system disorders) | 2 | 1 | 6
Encephalopathy (Nervous system disorders) | 2 | 0 | 6
Extremity-lower (gait/walking) (General disorders) | 1 | 1 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Neutrophils (Investigations) | 1 | 2 | 6
Platelets (Investigations) | 1 | 0 | 6
GGT (Investigations) | 1 | 1 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 1 | 7
Infection w/ gr3-4 neut- lung (Infections and infestations) | 0 | 1 | 7
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 | 2 | 7
Infection Gr0-2 neut- skin (Infections and infestations) | 3 | 2 | 8
Infection-other (Infections and infestations) | 1 | 3 | 9
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 9
Hypotension (Vascular disorders) | 2 | 3 | 10
Infection Gr0-2 neut- lung (Infections and infestations) | 5 | 2 | 10
Fracture (Injury, poisoning and procedural complications) | 5 | 1 | 11
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 11
Hemoglobin (Blood and lymphatic system disorders) | 4 | 0 | 12
Infection w/ gr3-4 neut- skin (Infections and infestations) | 6 | 1 | 12
Colitis- infectious (e.g. C.diff) (Infections and infestations) | 1 | 2 | 13
Neuropathy-motor (Nervous system disorders) | 2 | 3 | 14
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 5 | 6 | 15
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 6 | 6 | 15
Vascular access-Thrombosis/embolism (Vascular disorders) | 8 | 2 | 15
Bilirubin (Investigations) | 1 | 4 | 16
Typhlitis (Gastrointestinal disorders) | 0 | 2 | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 7 | 18
Hypokalemia (Metabolism and nutrition disorders) | 8 | 5 | 22
Seizure (Nervous system disorders) | 6 | 6 | 22
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 1 | 25
Pancreatitis (Gastrointestinal disorders) | 3 | 9 | 26
AST- SGOT (Investigations) | 4 | 8 | 28
Allergic reaction (Immune system disorders) | 6 | 14 | 33
Amylase (Investigations) | 5 | 6 | 37
Hypertension (Vascular disorders) | 2 | 3 | 39
ALT- SGPT (Investigations) | 9 | 10 | 48
Lipase (Investigations) | 12 | 10 | 49
Thrombosis/thrombus/embolism (Vascular disorders) | 10 | 12 | 55
Hypertriglyceridemia (Metabolism and nutrition disorders) | 12 | 20 | 69
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 15 | 21 | 100
Infection Gr 0-2 neut- blood (Infections and infestations) | 33 | 30 | 103
Infection w/ gr 3-4 neut- blood (Infections and infestations) | 25 | 29 | 234
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intramuscular Native E Coli L-asparaginase (IM-EC) (N=231) | Intravenous PEG-asparaginase (IV-PEG) (N=232) | Overall (N=794)
Agitation (Psychiatric disorders) | 0 | 1 | 1
Allergy-other (Immune system disorders) | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest/thoracic pain NOS (General disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Creatinine (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Infection Gr0-2 neut- bladder (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- bronchus (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- external ear (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut- eye NOS (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut- kidney (Infections and infestations) | 0 | 1 | 1
Infection Gr0-2 neut- lung (Infections and infestations) | 0 | 1 | 1
Infection Gr0-2 neut- lymphatic (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut- meninges (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- bronchus (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- catheter relate (Infections and infestations) | 1 | 0 | 1
Infection w/ gr3-4 neut- eye NOS (Infections and infestations) | 0 | 1 | 1
Infection w/ gr3-4 neut- larynx (Infections and infestations) | 1 | 0 | 1
Infection w/ gr3-4 neut- middle ear (Infections and infestations) | 1 | 0 | 1
Infection w/ gr3-4 neut- peritoneal (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- pharynx (Infections and infestations) | 1 | 0 | 1
Infection w/ gr3-4 neut- urinary tract (Infections and infestations) | 0 | 0 | 1
Infection w/ gr3-4 neut- wound (Infections and infestations) | 0 | 1 | 1
Infection w/ unk ANC catheter related (Infections and infestations) | 1 | 0 | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 0 | 0 | 1
Infection w/ unk ANC wound (Infections and infestations) | 0 | 0 | 1
Lipase (Investigations) | 0 | 0 | 1
Muco/stomatitis (symptom) anus (Gastrointestinal disorders) | 0 | 0 | 1
Muscle- pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neurologic-other (Nervous system disorders) | 0 | 1 | 1
Neutrophils (Investigations) | 0 | 0 | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Oral cavity- pain (Gastrointestinal disorders) | 0 | 0 | 1
Perforation- stomach (Gastrointestinal disorders) | 0 | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 0 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Speech impairment (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 2
Infection Gr0-2 neut- conjunctiva (Infections and infestations) | 1 | 1 | 2
Infection Gr0-2 neut- middle ear (Infections and infestations) | 1 | 1 | 2
Infection Gr0-2 neut- mucosa (Infections and infestations) | 0 | 0 | 2
Infection Gr0-2 neut- ungual (Infections and infestations) | 0 | 0 | 2
Infection Gr0-2 neut- upper airway (Infections and infestations) | 0 | 0 | 2
Infection Gr0-2 neut- wound (Infections and infestations) | 1 | 0 | 2
Infection w/ unk ANC lung (Infections and infestations) | 0 | 0 | 2
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 1 | 2
Joint- pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Personality (Psychiatric disorders) | 1 | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Ulcer- anus (Gastrointestinal disorders) | 0 | 0 | 2
Bone- pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Infection Gr0-2 neut- nose (Infections and infestations) | 2 | 0 | 3
Infection Gr0-2 neut- sinus (Infections and infestations) | 0 | 1 | 3
Infection Gr0-2 neut- skin (Infections and infestations) | 1 | 1 | 3
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 0 | 1 | 3
Infection w/ gr 3-4 neut- blood (Infections and infestations) | 0 | 1 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 3
Otitis- middle ear (non-infectious) (Ear and labyrinth disorders) | 0 | 3 | 3
ALT- SGPT (Investigations) | 1 | 0 | 4
Amylase (Investigations) | 1 | 2 | 4
CNS- hemorrhage (Nervous system disorders) | 4 | 0 | 4
Colitis (Gastrointestinal disorders) | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 4
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Infection Gr0-2 neut- oral cavity (Infections and infestations) | 0 | 2 | 4
Infection-other (Infections and infestations) | 2 | 0 | 4
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 4
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 4
Fever w/o neutropenia (General disorders) | 1 | 4 | 5
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 1 | 5
Neuropathy-motor (Nervous system disorders) | 0 | 0 | 5
Pain-other (General disorders) | 1 | 1 | 5
Skin-other (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
AST- SGOT (Investigations) | 2 | 0 | 6
Colitis- infectious (e.g. C.diff) (Infections and infestations) | 1 | 1 | 6
Vascular access-Thrombosis/embolism (Vascular disorders) | 1 | 3 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 7
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 5 | 1 | 10
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 7 | 14
Seizure (Nervous system disorders) | 5 | 5 | 17
Thrombosis/thrombus/embolism (Vascular disorders) | 9 | 4 | 22
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 7 | 7 | 31
Infection Gr 0-2 neut- blood (Infections and infestations) | 12 | 9 | 32
Allergic reaction (Immune system disorders) | 8 | 13 | 33
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 15 | 15 | 45
Hypertension (Vascular disorders) | 8 | 4 | 58
Pancreatitis (Gastrointestinal disorders) | 15 | 17 | 61
Fracture (Injury, poisoning and procedural complications) | 37 | 38 | 118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No